CLINICAL TRIAL: NCT01770665
Title: Mayo Clinic Validation of the MiCK Assay
Brief Title: Validation of the MiCK Assay
Acronym: MiCK Assay
Status: Terminated | Type: Observational
Why Stopped: Assay being revised and re-validated.
Sponsor: Pierian Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: MAYO1000
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Mesothelioma, Small Cell Lung Cancer, NSCLC
MeSH Terms: conditions — Mesothelioma; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Human cancerous tumor.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Mesothelioma
- all cancer types

SUMMARY:
Testing Mayo Clinic cancer patients with the results being correlated with prior patient therapy, performance status, and extent of disease.

DETAILED DESCRIPTION:
This study will be conducted in two phases.

During the Feasibility Phase, specimens from any tumor will be sent to the central DiaTech MiCK assay laboratory to determine the ease of sample acquisition, processing, transport, and assay interpretation.

Once DiaTech has completed analyses for the feasibility phase specimens and has confirmed that the sample acquisition, processing, transport, and assay interpretation are appropriate, we will proceed with the Demonstration Phase.

During the Mesothelioma Demonstration Phase, 20 mesothelioma samples will be assayed and the results will be correlated with prior patient therapy, performance status, and extent of disease.

ELIGIBILITY:
Inclusion Criteria:

* 20 subjects diagnosed with mesothelioma and 10 diagnosed with any malignancy.

Exclusion Criteria:

* patients that a sample cannot obtained for testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 subjects diagnosed with mesothelioma and 10 diagnosed with any malignancy.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Complete response and survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mary Karaus, Study Director — Mayo Clinic
Locations (1):
- Mayo Validation Support Services 3050 Superior Drive NW, Rochester, Minnesota, United States